CLINICAL TRIAL: NCT00001721
Title: Clinical and Basic Investigations Into Smith-Lemli-Opitz Syndrome
Brief Title: Study of Smith-Lemli-Opitz Syndrome
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 980081; 98-CH-0081
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-11-14

CONDITIONS: Smith-Lemli-Opitz Syndrome
Keywords: Cleft Palate; Cholesterol; Smith-Lemli-Opitz Syndrome (SLO)
MeSH Terms: conditions — Smith-Lemli-Opitz Syndrome; Cleft Palate | interventions — Cholesterol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients diagnosed with SLOS
  Interventions: Drug: Cholesterol Suspension; Drug: CRH; Drug: Cholesterol

INTERVENTIONS:
Drug: Cholesterol Suspension
Drug: CRH
Drug: Cholesterol

SUMMARY:
Smith-Lemli-Opitz Syndrome (SLOS) is a genetic disorder (autosomal recessive) caused by an abnormality in the production of cholesterol. The disorder can occur in both a "mild" or "severe" form. SLOS is associated with multiple birth defects and mental retardation. Some of the birth defects include; abnormal facial features, poor muscle tone, poor growth, shortened life span, and abnormalities of the heart, lungs, brain, gastrointestinal tract, limbs, genitalia, and kidneys.

There is no known cure for SLOS but recently patients have been treated with increased amounts of cholesterol in their diet. The cholesterol in a persons diet is unable to correct the abnormalities in the patient's organs, but researchers hope it will improve growth failure and mental retardation.

This study was developed to answer questions about the causes and complications of SLOS, as well as the effectiveness of cholesterol treatment. The study will enroll patients diagnosed with SLOS, and their mothers. The objectives of the study will be to address the following questions:

1. <TAB> What is the prognosis / natural history of the demyelination in the nervous system of patients with SLOS?
2. <TAB> Do patients with SLOS have other problems concerning the function of their endocrine systems?
3. <TAB>What are the genetic make-ups of patients with SLOS?
4. <TAB>Can further studies of cholesterol metabolism and genetic testing, using SLOS fibroblasts, increase the understanding of SLOS?<TAB>

DETAILED DESCRIPTION:
Smith-Lemli-Opitz syndrome (SLOS) is an autosomal recessive multiple congenital anomaly/mental retardation syndrome. Typical clinical features include a distinctive facial appearance, mental retardation, autistic behavior, hypotonia, failure to feed, poor growth, decreased life span, and variable structural anomalies of the heart, lungs, brain, gastrointestinal tract, limbs, genitalia and kidneys. The SLOS phenotypic spectrum is broad and variable. At the severe end of the spectrum SLOS is a lethal disorder with multiple major congenital anomalies; whereas, mild cases of SLOS present with a combination of minor physical stigmata, behavioral problems, and learning disabilities. SLOS is due to an inborn error of cholesterol biosynthesis. Biochemically, SLOS patients have a deficiency of 3beta-hydroxysterol delta(7)-reductase activity. 3beta-hydroxysterol delta(7)-reductase is an NADPH dependent microsomal enzyme that catalyzes the reduction of the C7(8) double bond of 7-dehydrocholesterol (7-DHC) to yield cholesterol in the last step of cholesterol biosynthesis via the Kandutsch-Russel pathway. This inborn error of cholesterol biosynthesis results in elevated tissue and serum 7-DHC levels and typically decreased serum and tissue cholesterol levels. In 1998 we established that the deficiency in 3beta-hydroxysterol delta(7)-reductase activity is due to mutation of the 3beta-hydroxysterol delta(7)-reductase gene (DHCR7). Once the biochemical defect in SLOS was identified, dietary cholesterol supplementation was proposed and employed as a therapeutic approach. Although developmental malformations remain fixed, dietary cholesterol supplementation appears to improve the overall health of these patients, and initial results have shown that dietary cholesterol supplementation has had a positive impact on some of the behavioral manifestations of this disorder. Although our understanding of this disorder has advanced over the last few years, many questions remain concerning the effectiveness of cholesterol replacement therapy, the long term prognosis for individuals on dietary cholesterol supplementation, and the need for adjunctive measures in the clinical management of SLOS patients. We propose to answer some of these questions by continuing our longitudinal natural history/prognosis study on patients with SLOS. We also plan on studying very closely related disorders such as lathosterolosis under this protocol. Lathosterolosis is caused by a deficiency in the enzyme sterol 3-beta-hydroxysteroid-delta-5-desaturase which is necessary for the conversion of lathosterol into 7-DHC. The clinical picture is very similar to SLOS with prominent features including microcephaly, ptosis bilateral 2,3 toe syndactyly. Lathosterolosis is also inherited in an autosomal recessive manner. Lethosterolosis is extremely rare with only 4 cases described in the literature so far and an estimated incidence of less than 1 in a million. The below objectives, protocol evaluations, risks, benefits and other pertinent issues apply to SLOS and lathosterolosis even if lathosterolosis is not explicitly named.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Any patient with biochemically confirmed SLOS will be accepted into this study. Patients of any age, either gender, or any ethnicity will be accepted into this study. No exclusions will be made based on race or gender. Historically, more males than females have been diagnosed as having SLOS. This bias was likely a result of the fact that genital hypoplasia is readily apparent in a male, and therefore the clinical diagnosis is easier to make in a male patient. SLOS syndrome appears more commonly in individuals of Northern European ancestry. Out of 150 biochemically proven cases, only one was an African American and no patients of Asian descent were reported. One SLOS mutant allele (R404C) appears to be present in individuals of French Canadian and Creole heritage. This likely represents a founder effect. One puzzling finding is that the carrier rate of the most common SLOS mutant allele in Black Canadians from Ontario and African Americans from Pennsylvania appears to be approximately 0.7%. However, clinical cases appear to be rare. The predominance of Caucasians reported in the literature may represent a bias of ascertainment of the disorder, variable presentation in different ethnic groups, or a founder effect in some ethnic groups. Because we function as a referral center with respect to recruitment, the ethnic background of our population is likely going to reflect the overall population of diagnosed cases.

EXCLUSION CRITERIA:

* Patients will be excluded if they cannot travel to the NIH because of their medical condition.
* Pregnant women will be excluded, and a negative urine pregnancy test will be required of menstruating women. This protocol focuses on biosampling. Increasing blood draws during pregnancy for research is not appropriate. Fetuses will be excluded since the proposed evaluations are not possible during fetal life.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with SLOS and other cholesterol disorders.
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 1998-09-13 (Actual)

PRIMARY OUTCOMES:
Neurocognitive Evalustion | Yearly
  Stabilization

CONTACTS AND LOCATIONS:
Overall Officials: Forbes D Porter, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Elias ER, Irons MB, Hurley AD, Tint GS, Salen G. Clinical effects of cholesterol supplementation in six patients with the Smith-Lemli-Opitz syndrome (SLOS). Am J Med Genet. 1997 Jan 31;68(3):305-10. doi: 10.1002/(sici)1096-8628(19970131)68:33.0.co;2-x. PMID 9024564
- [Background] Irons M, Elias ER, Abuelo D, Bull MJ, Greene CL, Johnson VP, Keppen L, Schanen C, Tint GS, Salen G. Treatment of Smith-Lemli-Opitz syndrome: results of a multicenter trial. Am J Med Genet. 1997 Jan 31;68(3):311-4. PMID 9024565
- [Background] Opitz JM. RSH/SLO ("Smith-Lemli-Opitz") syndrome: historical, genetic, and developmental considerations. Am J Med Genet. 1994 May 1;50(4):344-6. doi: 10.1002/ajmg.1320500408. PMID 8209912
- [Derived] Selvaraman A, Rahhal S, Bianconi S, Furnary T, Porter FD. Assessing Postnatal Mortality in Smith-Lemli-Opitz Syndrome. Am J Med Genet A. 2025 Feb;197(2):e63875. doi: 10.1002/ajmg.a.63875. Epub 2024 Sep 13. PMID 39271956
- [Derived] Campbell K, Cawley NX, Luke R, Scott KEJ, Johnson N, Farhat NY, Alexander D, Wassif CA, Li W, Cologna SM, Berry-Kravis E, Do AD, Dale RK, Porter FD. Identification of cerebral spinal fluid protein biomarkers in Niemann-Pick disease, type C1. Biomark Res. 2023 Jan 31;11(1):14. doi: 10.1186/s40364-023-00448-x. PMID 36721240
- [Derived] Thurm A, Tierney E, Farmer C, Albert P, Joseph L, Swedo S, Bianconi S, Bukelis I, Wheeler C, Sarphare G, Lanham D, Wassif CA, Porter FD. Development, behavior, and biomarker characterization of Smith-Lemli-Opitz syndrome: an update. J Neurodev Disord. 2016 Apr 5;8:12. doi: 10.1186/s11689-016-9145-x. eCollection 2016. PMID 27053961
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1998-CH-0081.html